CLINICAL TRIAL: NCT05239039
Title: Multi-centre, Open-label, Expanded Access Program of 900mg Intravenous (i.v.) Spesolimab in Patients With Generalized Pustular Psoriasis (GPP) Presenting With a Flare
Brief Title: An Expanded Access Program in China to Provide Spesolimab to People With a Flare-up in Generalized Pustular Psoriasis Who Have no Other Treatment Options
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0077
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spesolimab single dose treatment (Experimental): Patients with Generalized Pustular Psoriasis (GPP) presenting a flare received a single intravenous dose of 900 milligrams of spesolimab.
  Interventions: Drug: spesolimab
- Spesolimab double dose treatment (Experimental): Patients with Generalized Pustular Psoriasis (GPP) presenting a flare received a single intravenous dose of 900 milligrams of spesolimab. One week after the initial dose, patients received a second intravenous single dose of 900 mg of spesolimab due to persistence of flare symptoms.
  Interventions: Drug: spesolimab

INTERVENTIONS:
Drug: spesolimab — spesolimab

SUMMARY:
This Expanded Access Program in China is open to people with a serious skin disease called Generalized Pustular Psoriasis (GPP). This program provides a medicine called spesolimab to people with a GPP flare-up who have no alternative treatment options. This means that no therapy exists and participation in a clinical study is not possible.

Participants get a single infusion of spesolimab into a vein. They can get another spesolimab infusion one week after the first infusion if the doctors think it is helpful.

Participants are in the program for about 4 months and visit the study site about 5 times. Participants who benefit from the treatment during that time may repeat the treatment in case they experience a new GPP flare-up. The doctors regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of Generalized Pustular Psoriasis (GPP), consistent with European Rare and Severe Psoriasis Expert Network (ERASPEN) criteria, defined as primary, sterile, macroscopically visible pustules on non-acral skin (excluding cases where pustulation is restricted to psoriatic plaques). GPP can occur with or without systemic inflammation, with or without plaque-type psoriasis, and be either relapsing (>1 episode) or persistent (>3 months).
* Patient is experiencing a flare, defined as new or worsening of widespread eruption of sterile macroscopically visible pustules, with or without systemic inflammation, as assessed by the treating physician.
* Male or female patients, aged 18 to 75 years at time of enrolment. Women of childbearing potential (WOCBP) must be willing and able to use a highly effective method of birth control per International Council for Harmonization (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Signed and dated written informed consent in accordance with International Council for Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the program.
* No satisfactory authorized alternative therapy exists, as assessed by the treating physician.

Exclusion criteria

* Women who are pregnant, nursing, or who plan to become pregnant while in the program.

  -- Women who stop nursing before study drug administration do not need to be excluded from participating; they should refrain from breastfeeding for 16 weeks after the last spesolimab infusion.
* Severe, progressive, or uncontrolled hepatic disease, defined as >3-fold Upper Limit of Normal (ULN) elevation in Aspartate Transaminase (AST) or Alanine Aminotransferase (ALT) or alkaline phosphatase, or >2-fold ULN elevation in total bilirubin.
* Active systemic infections (fungal and bacterial disease) during the last 2 weeks prior to drug administration, as assessed by the treating physician.
* Increased risk of infectious complications (e.g. recent pyogenic infection, any congenital or acquired immunodeficiency (e.g. Human Immunodeficiency Virus (HIV)), past organ or stem cell transplantation), as assessed by the treating physician.
* Relevant chronic or acute infections, including active tuberculosis (TB), HIV infection or viral hepatitis at the time of drug administration.

  * Patients should be evaluated for TB infection prior to initiating treatment with spesolimab.
  * Anti-TB therapy should be considered, in accordance with local guidelines, prior to initiating spesolimab in patients with latent TB or a history of TB.
* History of allergy / hypersensitivity to systemically administered spesolimab or its excipients.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Immediate life-threatening flare of GPP requiring intensive care treatment according to the investigator's judgement. Life-threatening complications include cardiovascular / cytokine driven shock, pulmonary distress syndrome, or renal failure.

Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing Friendship Hospital, Beijing
  - West China Hospital, Chengdu
  - Southern Medical University Dermatology Hospital, Guangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Hangzhou Third People's Hospital, Hangzhou
  - Shandong Provincial Hospital of Dermatology, Jinan
  - Dermatology Hospital, Chinese Academy of Medical Sciences, Nanjing
  - Shanghai Skin Disease Hospital, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, multi-centre, single-arm trial, designed to provide early spesolimab to patients with Generalized Pustular Psoriasis (GPP) presenting with a flare and for whom no satisfactory authorised alternative therapy exists and who are unable to participate in a clinical trial, as assessed by the treating physician.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the project at any time for any reason given. Close monitoring of all subjects was adhered to throughout the expanded access program (EAP) conduct.
Period: Overall Study
Arm/Group | Spesolimab Single Dose Treatment | Spesolimab Double Dose Treatment
Started | 24 | 15
Completed | 24 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set: all patients who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Spesolimab Single Dose Treatment | Spesolimab Double Dose Treatment | Total
Number analyzed (Participants) | 24 | 15 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (14.7) | 38.3 (15.0) | 39.3 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 10 | 6 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 24 | 15 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 24 | 15 | 39

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Treatment Emergent Adverse Events (AEs)
Description: This outcome measured the number of patients with any treatment-emergent adverse event (AE). Treatment-emergent AEs are untoward medical events that appear or worsen during treatment.
Time Frame: From initial drug administration to: end of study treatment + residual effect period or end of study visit. Up to 16 weeks for the single dose group and up to 17 weeks for the double dose group.
Population: Treated set: all patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab Single Dose Treatment | Spesolimab Double Dose Treatment
Number analyzed (Participants) | 24 | 15
Participants | 18 | 12

2. Secondary Outcome: Occurrence of Treatment Emergent Serious Adverse Events (SAEs)
Description: This outcome measured the number of patients with serious adverse events (SAEs). SAEs are untoward medical occurrences that result in death, are life threatening, require inpatient hospitalisation, require prolongation of existing hospitalisation, result in persistent or significant disability/incapacity, result in a congenital anomaly/birth defect, or are deemed serious for any other medically important reason.
Time Frame: as for outcome 1
Population: Treated set: all patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab Single Dose Treatment | Spesolimab Double Dose Treatment
Number analyzed (Participants) | 24 | 15
Participants | 1 | 2

3. Secondary Outcome: Occurrence of Treatment Emergent Adverse Events of Special Interest (AESIs)
Description: This outcome measured the number of patients with any treatment-emergent adverse event of special interest (AESIs). AESIs relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this program. Potential severe DILIs (drug-induced liver injury), systemic hypersensitivity reactions, severe infections, opportunistic and mycobacterium tuberculosis infections, and peripheral neuropathy were considered as AESIs.
Time Frame: as for outcome 1
Population: Treated set: all patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab Single Dose Treatment | Spesolimab Double Dose Treatment
Number analyzed (Participants) | 24 | 15
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: From initial drug administration to: end of study treatment + residual effect period or end of study visit. Up to 16 weeks for the single dose group and up to 17 weeks for the double dose group.
Description: Treated set: all patients who received at least one dose of study drug.
Arm/Group | Spesolimab Single Dose Treatment | Spesolimab Double Dose Treatment
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/24 | 2/15
Other Adverse Events (participants affected / at risk) | 15/24 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab Single Dose Treatment (N=24) | Spesolimab Double Dose Treatment (N=15)
COVID-19 (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab Single Dose Treatment (N=24) | Spesolimab Double Dose Treatment (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 3
COVID-19 (Infections and infestations) | 3 | 6
Myringitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Tinea versicolour (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Blood albumin decreased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Prealbumin decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT05239039/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT05239039/SAP_001.pdf